CLINICAL TRIAL: NCT06899347
Title: Impact of PROphylactic Central COMpArtment Neck Dissection for 2-4 Cm Papillary Thyroid Carcinoma
Brief Title: The Role of Prophylactic Central Compartment Neck Dissection in the Management of 2 to 4 Cm Papillary Thyroid Carcinoma
Acronym: PRO-COMAND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leonardo Rossi (Other)
Responsible Party: Sponsor-Investigator, Leonardo Rossi, Senior Researcher in General Surgery, University of Pisa
Organization: University of Pisa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27092_MATERAZZI
Record Dates: First submitted 2025-03-13; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Papillary Thyroid Carcinoma; Central Compartment Neck Dissction; Thyroidectomy
Keywords: papillary thyroid carcinoma; prophylactic central compartment neck dissection; thyroidectomy; surgical complications; outcomes
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total Thyroidectomy (No Intervention)
- Total Thyroidectomy + pCCND (Experimental)
  Interventions: Procedure: Total Thyroidectomy + Central Compartment Neck Dissection

INTERVENTIONS:
Procedure: Total Thyroidectomy + Central Compartment Neck Dissection — Thyroidectomy will be performed with the patient in the supine position with the neck hyperextended. A 3 to 6 cm transverse cervicotomy, two fingers above the sternal notch, will be performed, and the midline will be opened. After the inferior laryngeal nerve and parathyroids are visualized, the thyroidectomy will be achieved.
  When performed, pCCND will aim at removing the nodes of Level VI, which has been reported to contain the thyroid gland and the adjacent nodes bordered superiorly by the hyoid bone, inferiorly by the brachiocephalic artery, and laterally on each side by the carotid sheaths
  Arms: Total Thyroidectomy + pCCND

SUMMARY:
This randomized prospective study aims to evaluate the advantages and disadvantages (both oncologic and surgical) of prophylactic central compartment neck dissection for clinically node-negative 2-4 cm papillary thyroid carcinoma patients who have been treated either with total thyroidectomy alone or with total thyroidectomy + prophylactic central compartment neck dissection .

ELIGIBILITY:
Inclusion Criteria:

1. PTC documented by fine needle aspiration cytology (FNAC) (TIR 4 or TIR 5 according to the Italian consensus for the classification and reporting of thyroid cytology [15]);
2. no pre-operative evidence of lymph node metastases (cN0) at palpation and neck ultrasound (US);
3. no clinical evidence of distant metastasis at diagnosis;
4. age ≥ 18 years.

Exclusion Criteria:

1. histotypes other than PTC;
2. evidence of lymph node metastases during surgery even if not previously diagnosed;
3. presence of distant metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Persistent or Recurrent Papillary Thyroid Carcinoma | from enrollment to 1, 3, 5 and 10 years
  Persistent or recurrent disease refers to the presence or reappearance of cancerous tissue despite initial treatment. It is assessed through a combination of biochemical and imaging studies. Biochemically, elevated serum thyroglobulin (Tg) or detectable anti-thyroglobulin antibodies (TgAb) after total thyroidectomy may suggest residual or recurrent disease. Moreover, they may represent a biochemical incomplete or indeterminate response to therapy. On the other hand, imaging techniques such as neck ultrasound or CT scan can identify structural disease.
Overall Survival | from the enrollment to 1, 3, 5, and 10 years
  Overall survival is the most comprehensive indicator of treatment efficacy and patient prognosis. It is typically assessed through survival analysis methods, such as Kaplan-Meier curves, and is expressed as a percentage of patients alive at specific time points.

SECONDARY OUTCOMES:
Surgical Complications | from enrollment to 1, 3, 5 and 10 years
  Complications following thyroidectomy are mainly hypoparathyroidism, vocal cord palsy and bleeding. They are assessed through clinical evaluation, laboratory tests (e.g., calcium and PTH levels for hypoparathyroidism), and laryngoscopy and / or transcutaneous laryngeal ultrasound for vocal cord function.

IPD SHARING:
Plan to Share IPD: Undecided